CLINICAL TRIAL: NCT06377956
Title: Associations Between Gut Length, Gut Microbiota and Food Assimilation Efficiency of Healthy Individuals
Brief Title: The Associations Between Gut Length, Gut Microbiota and Food Assimilation
Status: Completed | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, chief researcher, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-240415-H0717
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Nutrition; Food Preferences; Metabolic Syndrome, Protection Against
Keywords: Metabolism; Microbiome/microbiota; Body composition; Food intake; Food preference
MeSH Terms: conditions — Food Preferences; Metabolic Syndrome | interventions — Observation; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age between 18-40 years old, 100subjects（50 female and 50 man）: He Shuang(Polyethylene Glycol Electrolytes Powder):1/1.5 sachets of PEG(68.56-102.84g dissolved in water with1/1.5L ) were provided to volunteers based on body weight(BW): BW<60 kg, 1 sachet , BW≥60 kg, 1.5 sachets, drinking an average of 200/250 mL every 15 minutes. It will cause frequent bowel motions or diarrhoea for a couple of hours afterwards.
  Raceanisodamine Hydrochloride Injection: intramuscular injection of Raceanisodamine Hydrochloride Injection with 10mg. It may cause dry mouth, red face and blurred vision. The half-life of the medicine is 40 minutes and most of the above symptoms disappear within 1 to 3 hours.
  Interventions: Other: Observation without intervention

INTERVENTIONS:
Other: Observation without intervention — Observation of gut length, food intake, fecal and urine calories, body composition, microbiota, metabolic rate, metabolomics.

SUMMARY:
The purpose of this observational study is to explore the relationships between gut length, the microbiota and food energy assimilation rates in humans.

DETAILED DESCRIPTION:
The focus of this work is to characterize the relationship between gut length, gut microbiota and food energy assimilation rate in healthy individuals.

The gut will be scanned using Magnetic Resonance Imaging (MRI) to calculate gut length. To obtain clearer images, volunteers will be asked to drink 1/1.5 sachet of He Shuang (polyethylene glycol electrolyte powder, molecular weight of 4000) and injected Raceanisodamine Hydrochloride Injection with 10 mg by intramuscular. Volunteers will be asked to drink He Shuang, which dissolved in 1/1.5L of water for the purpose of filling the intestines. As a contrast to improve imaging during scanning.

Volunteers will be given the experimental meal, which providing enough energy for volunteers to eat as much as they want. Feces and urine will be collected to calculate the assimilation rate. To more accurately label the food, edible polyethylene glycol with a molecular weight of 3350(PEG3350) is used. Provides 1.5g of PEG3350 per day, to be used with meals. PEG3350 reaches a steady state in the intestinal tract for 3 days. Food will be provided for seven days during the test period, the first three days are aimed at stabilizing the PEG3350 in the intestine, and the samples to be counted are mainly collected in the last four days. Food assimilation rate and metabolizable energy will be calculated for the 4-day.

The gut microbiota will be analyzed by metagenomics and metabolomics. This study combines metabolomics analysis techniques with imaging and physiological measurements to focus on the potential relationship between gut length and food absorption rates. Researchers anticipate recruiting up to 100 healthy volunteers (body mass index ≥ 18.5).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years old, healthy and disease free.
* Regular bowel movements.

Exclusion Criteria:

* Individuals who are constipated or suffer from intestinal disorders;
* Individuals with mental illnesses such as depression and claustrophobia;
* Individuals with glaucoma and prostate hypertrophy;
* Metal implants in the body;
* Pregnant and lactating women;
* Individuals with blood phobia, pathologic hypotension or hypertension;
* Use of antibiotics, probiotics, oral laxatives within 8 weeks;
* Individuals with metabolic diseases (e.g., chronic diseases such as diabetes mellitus); recent weight loss due to various medical reasons;
* Individuals with infectious diseases (e.g. HIV);
* Irregular diet, lifestyle, addiction to tobacco, alcohol or drugs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 individuals, 50 female and 50 male
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Gut length | Through study completion for one year, will be measured on arrival.
  Volunteers will be scanned Magnetic Resonance Imaging(Shanghai united imaging, uMR 790).
Energy intake | Through study completion for one year, will be measured on arrival.
  Response on standard feeding table, the food consumption will be recorded continuously by balances underneath each food dish. The total energy intake will be calculated in KJ (kilojoule).
Fecal energy | Through study completion for one year, will be measured on arrival
  Measuring the heat produced by burning dried feces using an oxygen bomb calorimeter (Parr6400). The total energy per gram tissue will be calculated in kJ (kilojoule)/g.
Microbiome/Microbiota | Through study completion for one year, will be measured on arrival.
  Abundance of gut microbiome will be from Metagenomic profiling of feces by Illumina.
Metabolites | Through study completion for one year, will be measured on arrival.
  Abundance of metabolites will be from metabolomic profiling of feces by LC-MS (liquid chromatography mass spectrometry).

SECONDARY OUTCOMES:
Urine energy content | Through study completion for one year, will be measured on arrival.
  Energy content will be evaluated by measuring the heat energy produced when burning dried urine using an oxygen bomb calorimeter (Parr6400). The total energy per gram tissue will be calculated in kJ (kilojoule)/g.
Body weight | Through study completion for one year, will be measured on arrival.
  Volunteers will be asked to fast for 10 hours and measured fasting weight.
Waist circumferences | Through study completion for one year, will be measured on arrival.
  Waist circumferences will be measured using a whole body laser scanner(TG2000-F).
Height | Through study completion for one year, will be measured on arrival.
  Height will be measured by seca 217 stable stadiometer.
Bone mass | Through study completion for one year, will be measured on arrival.
  Bone mass will be measured by Dual Energy X-ray Absorptiometry (Horizon Wi).
Hip circumferences | Through study completion for one year, will be measured on arrival.
  Hip circumferences will be measured using a whole body laser scanner(TG2000-F).
Fat free mass | Through study completion for one year, will be measured on arrival.
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, MC-980) and BOD POD(COS MED,BOD POD 2020).
Heart rate | Through study completion for one year, will be measured on arrival.
  Heart rate will be measured using an Omron sphygmomanometer.
Resting energy expenditure | Through study completion for one year, will be measured on arrival.
  The measurement of resting energy expenditure will be performed using indirect calorimetry(Whole room calorimetry) for 24h.
Thermic effect of food | Through study completion for one year, will be measured on arrival.
  The measurement of resting energy expenditure will be performed using indirect calorimetry(Whole room calorimetry) for 24h.
Body shape | Through study completion for one year, will be measured on arrival.
  Body shape will be measured using a whole body laser scanner(TG2000-F)
Fat mass | Through study completion for one year, will be measured on arrival.
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ) and BOD POD(COS MED,BOD POD 2020).
Blood pressure | Through study completion for one year, will be measured on arrival.
  Systolic and diastolic blood pressure will be measured using an Omron sphygmomanometer.
Total daily water volume | Through study completion for one year, will be measured on arrival.
  Calculate the total amount of water to be consumed in a day by providing water cups with a graduated scale.
Physical activity | Through study completion for one year, will be measured on arrival.
  Physical activity of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 7 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day where the wear time is less than 12 hours. For a valid measure the goal is to get 2 weekday and 2 weekend days.
Bristol Stool Scale | Through study completion for one year, will be measured on arrival.
  Scoring of stool forms according to the Bristol Stool Scale, whice classified according to faecal characteristics. It has seven types. Types 1 and 2 indicate the presence of constipation, types 3 and 4 are ideal stool shapes, and types 5 to 7 represent possible diarrhoea.
Total daily urine volume | Through study completion for one year, will be measured on arrival.
  Collect the urine sample within a day in a graduated container.
Gut transit time | Through study completion for one year, will be measured on arrival.
  Recording the time of intake of food-grade blue pigment and the time of excretion
Food macronutrient content | Through study completion for one year, will be measured on arrival.
  Detection of carbohydrates, proteins and fats in food by chemical analysis.
Feces macronutrient content | Through study completion for one year, will be measured on arrival.
  Detection of carbohydrates, proteins and fats in feces by chemical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Study Chair — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No